CLINICAL TRIAL: NCT06976983
Title: Effects of Transcranial Static Magnetic Stimulation (tSMS) in the Treatment of Hyperkinetic Symptoms of Huntington's Disease
Brief Title: Transcranial Static Magnetic Stimulation (tSMS) in Huntington's Disease (HD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Diego Centonze, MD, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD2024
Record Dates: First submitted 2024-11-14; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Huntington Disease
Keywords: huntington disease; transcranial stimulation with static magnetic field; hyperckinesia
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD patients undergo real tSMS (Active Comparator): Each HD patients undergo tSMS (real) in two sessions per day, each lasting 60 minutes.
  Interventions: Device: Portable ergonomic helmet for real tSMS
- HD patients undergo placebo tSMS (Sham Comparator): Each HD patients undergo tSMS (placebo), in two sessions per day, each lasting 60 minutes.
  Interventions: Device: portable ergonomic helmet for placebo tSMS

INTERVENTIONS:
Device: Portable ergonomic helmet for real tSMS — Unlike repetitive magnetic stimulation (rTMS), tSMS is attracting considerable interest because it is more manageable and easy to apply. It is a method applicable through a portable ergonomic helmet that shifts the paradigm of non-invasive brain stimulation (NIBS) from a center-based therapeutic model to a home-based one.
  Arms: HD patients undergo real tSMS
Device: portable ergonomic helmet for placebo tSMS — Unlike repetitive magnetic stimulation (rTMS), tSMS is attracting considerable interest because it is more manageable and easy to apply. It is a method applicable through a portable ergonomic helmet that shifts the paradigm of non-invasive brain stimulation (NIBS) from a center-based therapeutic model to a home-based one.
  Arms: HD patients undergo placebo tSMS

SUMMARY:
Huntington's disease (HD) is a neurodegenerative pathology characterized by choreic hyperkinesias which represent the typical motor symptom and are represented by involuntary, aimless, irregular, recurrent, unpredictable and non-rhythmic movements of the trunk, face and limbs.

Non-invasive brain neuromodulation has been proposed as a possible treatment for involuntary movements in several clinical conditions including HD.

The objective of the study is to evaluate the effect of home treatment with repeated sessions of transcranial static magnetic field stimulation (tSMS) in safely reducing choreic hyperkinesis in HD patients.

DETAILED DESCRIPTION:
A two-week course of repetitive magnetic stimulation (rTMS) has been shown to exert persistent clinical beneficial effects, reducing peak drug dyskinesias for up to four weeks after the end of the stimulation period. rTMS has also been reported to have a beneficial effect in HD. In particular, the stimulation showed a significant reduction in involuntary movements in a group of symptomatic patients.

Unlike rTMS, tSMS is attracting considerable interest because it is more manageable and easier to apply. This is a method applicable using a portable ergonomic helmet that shifts the paradigm of non-invasive brain stimulation (NIBS) from a center-based therapeutic model to a home-based one.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HD genetically confirmed (number of CAG triplets ≥36)
* Presence of chorea movements quantified with a score ≥ 10 on the sum of the scores of the subscale of the Unified Huntington's Disease Rating Scale (UHDRS) for the evaluation of maximum chorea for the facial, oro-bucco-lingual, truncal, four limbs districts
* Ability to provide written informed consent
* No changes in drug therapy in the 8 weeks prior to the baseline visit
* No changes in drug therapy for the entire duration of the study

Exclusion Criteria:

* Contraindications to exposure to magnetic fields
* Patients who are pregnant or breastfeeding
* Presence of significant risk of suicidal behavior
* Patients who have received an investigational drug in a clinical trial within 30 days of the baseline visit or have planned to use such an investigational drug during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of choreic hyperkinesias and akathisia in patients with HD | The project aims to evaluate the efficacy of tSMS in reducing choreic hyperkinesias in patients after 1 month stimulation
  The project aims to evaluate the efficacy of tSMS in reducing choreic hyperkinesias in 30 patients with HD. The Unified Huntington's Disease Rating Scale will be used to assessed maximal chorea in different body districts (face, bucco-oral-lingual, trunk, upper and lower extremity) before and after treatment. Akathisia will be instead determined with the Barnes Akathisia Rating Scale.

SECONDARY OUTCOMES:
Modulation of neuropsychiatric symptoms | The project aims to evaluate the efficacy of tSMS in reducing choreic hyperkinesias in patients after 1 month stimulation
  As a further objective, the project aims to evaluate the possible modulation of neuropsychiatric symptoms commonly associated with the disease by using the Beck Depression Inventory-II, State-Trait Anxiety Inventory and Columbia Suicide Severity Rating Scale.
  tSMS is a non-invasive method and almost free of adverse events if administered in well-selected patients. This method could represent a complement to pharmacological therapy in the advanced stages or, possibly, replace it in the early stages of the disease by reducing the potential side effects secondary to prolonged pharmacological treatment.

REFERENCES:
- [Background] Tan B, Shishegar R, Fornito A, Poudel G, Georgiou-Karistianis N. Longitudinal mapping of cortical surface changes in Huntington's Disease. Brain Imaging Behav. 2022 Jun;16(3):1381-1391. doi: 10.1007/s11682-021-00625-2. Epub 2022 Jan 14. PMID 35029800
- [Background] Stoker TB, Mason SL, Greenland JC, Holden ST, Santini H, Barker RA. Huntington's disease: diagnosis and management. Pract Neurol. 2022 Feb;22(1):32-41. doi: 10.1136/practneurol-2021-003074. Epub 2021 Aug 19. PMID 34413240
- [Background] Spargo E, Everall IP, Lantos PL. Neuronal loss in the hippocampus in Huntington's disease: a comparison with HIV infection. J Neurol Neurosurg Psychiatry. 1993 May;56(5):487-91. doi: 10.1136/jnnp.56.5.487. PMID 8505640
- [Background] Rubinsztein DC. How does the Huntington's disease mutation damage cells? Sci Aging Knowledge Environ. 2003 Sep 17;2003(37):PE26. doi: 10.1126/sageke.2003.37.pe26. PMID 13679594
- [Background] Quinn N, Schrag A. Huntington's disease and other choreas. J Neurol. 1998 Nov;245(11):709-16. doi: 10.1007/s004150050272. PMID 9808238
- [Background] Kremer HP, Roos RA, Dingjan GM, Bots GT, Bruyn GW, Hofman MA. The hypothalamic lateral tuberal nucleus and the characteristics of neuronal loss in Huntington's disease. Neurosci Lett. 1991 Oct 28;132(1):101-4. doi: 10.1016/0304-3940(91)90443-w. PMID 1838577
- [Background] Kremer B, Weber B, Hayden MR. New insights into the clinical features, pathogenesis and molecular genetics of Huntington disease. Brain Pathol. 1992 Oct;2(4):321-35. doi: 10.1111/j.1750-3639.1992.tb00709.x. PMID 1341966
- [Background] Jose L, Martins LB, Cordeiro TM, Lee K, Diaz AP, Ahn H, Teixeira AL. Non-Invasive Neuromodulation Methods to Alleviate Symptoms of Huntington's Disease: A Systematic Review of the Literature. J Clin Med. 2023 Mar 2;12(5):2002. doi: 10.3390/jcm12052002. PMID 36902788
- [Background] Jiang A, Handley RR, Lehnert K, Snell RG. From Pathogenesis to Therapeutics: A Review of 150 Years of Huntington's Disease Research. Int J Mol Sci. 2023 Aug 21;24(16):13021. doi: 10.3390/ijms241613021. PMID 37629202
- [Background] Hensel L, Ludtke J, Brouzou KO, Eickhoff SB, Kamp D, Schilbach L. Noninvasive brain stimulation in autism: review and outlook for personalized interventions in adult patients. Cereb Cortex. 2024 May 2;34(13):8-18. doi: 10.1093/cercor/bhae096. PMID 38696602
- [Background] Heinsen H, Rub U, Bauer M, Ulmar G, Bethke B, Schuler M, Bocker F, Eisenmenger W, Gotz M, Korr H, Schmitz C. Nerve cell loss in the thalamic mediodorsal nucleus in Huntington's disease. Acta Neuropathol. 1999 Jun;97(6):613-22. doi: 10.1007/s004010051037. PMID 10378380
- [Background] Dileone M, Ammann C, Catanzaro V, Pagge C, Piredda R, Monje MHG, Navalpotro-Gomez I, Bergareche A, Rodriguez-Oroz MC, Vela-Desojo L, Alonso-Frech F, Catalan MJ, Molina JA, Lopez-Ariztegu N, Oliviero A, Obeso JA, Foffani G. Home-based transcranial static magnetic field stimulation of the motor cortex for treating levodopa-induced dyskinesias in Parkinson's disease: A randomized controlled trial. Brain Stimul. 2022 May-Jun;15(3):857-860. doi: 10.1016/j.brs.2022.05.012. Epub 2022 May 21. No abstract available. PMID 35609815
- [Background] Cole E, O'Sullivan SJ, Tik M, Williams NR. Accelerated Theta Burst Stimulation: Safety, Efficacy, and Future Advancements. Biol Psychiatry. 2024 Mar 15;95(6):523-535. doi: 10.1016/j.biopsych.2023.12.004. PMID 38383091
- [Background] Calderon-Villalon J, Ramirez-Garcia G, Fernandez-Ruiz J, Sangri-Gil F, Campos-Romo A, Galvez V. Planning deficits in Huntington's disease: A brain structural correlation by voxel-based morphometry. PLoS One. 2021 Mar 24;16(3):e0249144. doi: 10.1371/journal.pone.0249144. eCollection 2021. PMID 33760890
- [Background] Caballero-Insaurriaga J, Pineda-Pardo JA, Obeso I, Oliviero A, Foffani G. Noninvasive modulation of human corticostriatal activity. Proc Natl Acad Sci U S A. 2023 Apr 11;120(15):e2219693120. doi: 10.1073/pnas.2219693120. Epub 2023 Apr 6. PMID 37023134
- [Background] Brusa L, Versace V, Koch G, Bernardi G, Iani C, Stanzione P, Centonze D. Improvement of choreic movements by 1 Hz repetitive transcranial magnetic stimulation in Huntington's disease patients. Ann Neurol. 2005 Oct;58(4):655-6. doi: 10.1002/ana.20613. No abstract available. PMID 16178020